CLINICAL TRIAL: NCT03115775
Title: Randomized Controlled Trial to Evaluate the Independent and Combined Effects of Conjugated Linoleic Acids and Vitamin D on Muscle Protein Turnover in Older Adults
Brief Title: CLA and Vitamin D on Protein Turnover
Acronym: TM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: BASF (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 201702113
Record Dates: First submitted 2017-04-07; First posted 2017-04-14 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Protein
MeSH Terms: interventions — Linoleic Acids, Conjugated; Vitamin D; Corn Oil

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conjugated linoleic acid (Tonalin) (Active Comparator): Conjugated linoleic acid (4000 mg Tonalin FFA 80 per day)
  Interventions: Dietary Supplement: Conjugated linoleic acid
- Vitamin D (Active Comparator): Vitamin D3 (2000 IU per day)
  Interventions: Dietary Supplement: Vitamin D
- Conjugated linoleic acid and Vitamin D (Active Comparator): Conjugated linoleic acid (4000 mg Tonalin FFA 80) and Vitamin D (2000 IU) per day
  Interventions: Dietary Supplement: Conjugated linoleic acid and Vitamin D
- Placebo (Placebo Comparator): Corn oil (4000 mg per day)
  Interventions: Other: Corn oil (placebo)

INTERVENTIONS:
Dietary Supplement: Conjugated linoleic acid — Intervention will last up to 8 weeks. Subjects will receive conjugated linoleic acid (4000 mg Tonalin FFA 80) daily.
  Other Names: Tonalin
  Arms: Conjugated linoleic acid (Tonalin)
Dietary Supplement: Vitamin D — Intervention will last up to 8 weeks. Subjects will receive vitamin D3 (2000 IU) daily.
  Arms: Vitamin D
Dietary Supplement: Conjugated linoleic acid and Vitamin D — Intervention will last up to 8 weeks. Subjects will receive conjugated linoleic acid (4000 mg Tonalin FFA 80) and vitamin D3 (2000 IU) daily.
  Arms: Conjugated linoleic acid and Vitamin D
Other: Corn oil (placebo) — Intervention will last up to 8 weeks. Subjects will receive corn oil (4000 mg) daily.
  Arms: Placebo

SUMMARY:
To conduct a randomized, double-blind, controlled clinical trial to determine the independent and combined effects of dietary conjugated linoleic acid (CLA) and vitamin D supplementation on anabolic signaling, the expression of growth regulatory factors, and muscle protein turnover in older adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/= 18.5 and </= 35.0
* Serum 25OH-VitD3 < 35 ng/ml

Exclusion Criteria:

* Diabetes
* COPD

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in post-absorptive muscle protein synthesis | Baseline and 8 weeks
  A stable isotope labelled amino acid infusion, in conjunction with blood and muscle tissue sampling and mathematical modelling analysis will be used to measure post-absorptive muscle protein synthesis.
Change in combined amino acid and insulin stimulated muscle protein synthesis | Baseline and 8 weeks
  A stable isotope labelled amino acid infusion, in conjunction with insulin and mixed amino acid infusion, blood and muscle tissue sampling and mathematical modelling analysis will be used to measure muscle protein synthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Vliet S, Fappi A, Reeds DN, Mittendorfer B. No independent or combined effects of vitamin D and conjugated linoleic acids on muscle protein synthesis in older adults: a randomized, double-blind, placebo-controlled clinical trial. Am J Clin Nutr. 2020 Nov 11;112(5):1382-1389. doi: 10.1093/ajcn/nqaa240. PMID 32860399